CLINICAL TRIAL: NCT06382298
Title: Health Effects of Cottonseed Oil Versus Matched Composition Diets in Humans
Brief Title: Cottonseed Oil Versus Matched PUFA Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Professor, Department Head of Kinesiology, Director of UGA Obesity Initiative, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PROJECT00009332
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Dyslipidemia; Overweight and Obesity; Nutrition, Healthy
MeSH Terms: conditions — Dyslipidemias; Overweight; Obesity | interventions — Cottonseed Oil

STUDY DESIGN:
Intervention Model Description: Three groups of 28-day parallel feeding trials with two groups receiving 20% of energy needs from CSO, or matched PUFA diet, and one group serving as control receiving 20% of energy needs as a mixture of oils that match the fatty acid profile of the average American intake.
Who Masked: Participant, Investigator
Masking Description: Participants are blinded to oil intervention group. Investigator blinded to participant's oil intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- COTTONSEED OIL (Experimental): Participants are given a daily shake enriched with cottonseed oil and instructed on how to substitute provided study shake into usual diet to maintain caloric balance.
  Interventions: Other: COTTONSEED OIL
- MATCHED PUFA DIET (Experimental): Participants are given a daily shake enriched with a mixture of oils with a similar fatty acid profile to CSO and instructed on how to substitute provided study shake into usual diet to maintain caloric balance.
  Interventions: Other: MATCHED PUFA DIET
- CONTROL (Active Comparator): Participants are given a daily shake enriched with a mixture of oils that match the fatty acid profile of the average American diet, and instructed on how to substitute provided study shake into usual diet to maintain caloric balance.
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: COTTONSEED OIL — Participants are provided a breakfast shake that meets 20% of participant's daily estimated energy needs as cottonseed oil for 28 days.
  Arms: COTTONSEED OIL
Other: MATCHED PUFA DIET — Participants are provided a breakfast shake that meets 20% of participant's daily estimated energy needs from oils with similar fatty acid composition as CSO for 28 days.
  Arms: MATCHED PUFA DIET
Other: CONTROL — Participants are provided a breakfast shake that meets 20% of participant's daily estimated energy needs as a mixture of oils that match the average American fat intake for 28 days.
  Arms: CONTROL

SUMMARY:
Cardiovascular disease risk factors, including higher BMIs and poor cholesterol profiles, are on the rise and contribute to the United States' growing disease burden. Cottonseed oil (CSO) is found readily in the food supply, and the investigator's previous studies have demonstrated that incorporating CSO into the diet is sufficient to improve fasting cholesterol profile and improve postprandial lipid and/or glycemic responses in both healthy, and at-risk populations. This study aims to compare CSO to a fatty acid composition-matched diet, on changes in fasting and postprandial lipid metabolism and markers of chronic disease risk.

The specific aims are:

* Examine the impact of CSO vs. PUFA on fasting and postprandial lipids.
* Examine the impact of CSO on other markers of chronic disease risk.

Participants will be asked to:

* Consume provided meal replacement shakes daily for 28-days.
* Attend three weekly short visits for fasting blood draws, body measurements, and collect the next week of study materials,
* Attend two longer (5.5h) testing visits which include eating a standardized breakfast meal and having blood drawn periodically before and after breakfast.

Researchers will compare CSO vs. PUFA and control groups (receiving a mixture of oils) to see if CSO is unique in imparting health benefits when compared with similar matched oil diets.

DETAILED DESCRIPTION:
Accounting for nearly 1 in every 4 deaths in the U.S., cardiovascular disease (CVD) is the leading cause of death for adults. One risk factor for CVD is hypercholesterolemia which can double the risk for this disease. Cottonseed oil is a rich source of poly-unsaturated fatty acids (PUFAs). Despite having a relatively high amount of saturated fatty acids, preliminary studies demonstrate that incorporating CSO into a diet is sufficient to reduce blood lipid profiles and select postprandial measures of metabolism. These improvements in lipid metabolism may be due to the general fatty acid (FA) composition of CSO; however, evidence shows that a fatty acid unique to CSO, dihydrosterculic acid (DHSA), may be responsible for some, if not all, the positive lipid lowering effects.

This prospective clinical study is a double-blinded, randomized control trial in adults at increased risk for cardiovascular disease (poor cholesterol profiles or overweight/obesity). There are three diet interventions: CSO (20% energy needs from CSO), matched-PUFA (20% energy needs from non-CSO matched PUFA sources), and Control (20% of energy needs from control oil mixture representative of the average fatty acid composition consumed by U.S. adults). The study protocol consists of a 28-day intervention where participants are provided breakfast shakes that contain a different oil, or mixture of oils, depending on the participant's random group assignment.

There are a total of 6 testing visits: screening (v0), pre-intervention (v1), 3 weekly short visits (v2, v3, v4), and post-intervention (v5).

At screening (v0), qualification is confirmed based on anthropometrics and fasting blood draw, which is analyzed for a cholesterol panel and blood glucose. Additionally, energy requirements are estimated at this visit for use in the diet intervention.

At v1, participants will have anthropometrics measured, including body composition by dual-energy x-ray absorptiometry (DXA). Fasting and postprandial blood draws for a 5h period will occur following a high saturated-fat meal challenge which delivers 35% of the participant's estimated energy needs.

28-day dietary intervention: Participants will consume a daily shake corresponding to the participant's randomly assigned group. The ingredients for the breakfast shakes are identical between groups, the only difference being the composition of assigned oil provided. The breakfast shakes are portioned based on individual energy needs as estimated at v0.

Participants return weekly (v2, v3, v4), to return study materials and collect shakes for the next week. At these weekly visits, participants also have a fasting blood draw, body measures, and consume the daily breakfast shake in the lab.

At the end of the 28-day dietary intervention, participants return for v5, where all procedures from v1 are repeated.

As decided a priori, we will complete a per protocol analysis.

The investigators hypothesize that CSO will improve the proposed overall health outcomes and markers of chronic disease risk when compared with the matched PUFA and control groups.

ELIGIBILITY:
Inclusion Criteria:

* 25-75 year-old men and women at increased risk for cardiovascular disease. Increased risk for cardiovascular disease will be defined by either elevated cholesterol profiles -or- overweight/obesity.
* Elevated cholesterol profiles will be defined as:

-"Borderline High" and/or "at risk" in two of more of the following variables (total cholesterol: 180-239 mg/dL, LDL cholesterol 110-159 mg/dL, triglycerides 130-199 mg/dL) --or--

* "High" in total cholesterol (240 mg/dL and higher), LDL (160 mg/dL or higher), or triglycerides (between 200-350 mg/dL).

Overweight/obesity will be defined by body mass index >25 kg/m².

Exclusion Criteria:

* Probable familial hypercholesterolemia, defined by: total cholesterol greater than 290 mg/dL or LDL levels greater than 190 mg/dL plus a family history of myocardial infarction (MI) before 50 years of age in a 2nd-degree relative or below age 60 in a 1st-degree relative.
* Women on hormone replacement therapy less than 2 years.
* Women who are pregnant
* individuals who regularly exercise more than 3h/w
* weight gain or loss of more than 5% body weight in the past 3 months
* plans to begin a weight loss/exercise regimen during the trial
* history of medical or surgical events that could affect digestion or swallowing
* gastrointestinal surgeries, conditions, or disorders
* any chronic diseases (including moderate to severe asthma, chronic lung disease, and kidney disease),
* metabolic disease
* atherosclerosis
* previous MI or stroke
* cancer
* fasting blood glucose levels greater than 126 mg/dL
* blood pressure greater than 180/120 mmHg
* medication use affecting digestion an absorption, metabolism (e.g. thyroid meds), lipid-lowering medications, medications for diabetes, steroid/hormone therapies, or current antibiotic cycles
* medically prescribed or special diets
* Food allergies (specific to the foods in the study, including wheat, dairy, and cottonseed oil)
* fish oil supplements
* excessive alcohol use (greater than 3 drinks/day for men; greater than 2 drinks/day for women)
* tobacco or nicotine use
* underweight BMI (<18.5 kg/m²)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in fasting serum lipoprotein and cholesterol concentrations | baseline, 4 weeks
  The concentration of fasting serum total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, apolipoprotein B (mg/dL)
Change in fasting and postprandial plasma triglyceride concentrations | baseline, 4 weeks
  The concentration of plasma triglycerides before and after the high saturated fat meal challenge at both pre-and post-intervention visits (mg/dL)
Change in fasting and postprandial plasma non-esterified fatty acid (NEFA) concentrations | baseline, 4 weeks
  The concentration of plasma NEFAs before and after the high saturated fat meal challenge at both pre- and post- intervention visits (mEq/L)
Change in fasting and postprandial plasma appetite control hormones concentrations | baseline, 4 weeks
  The concentration of plasma appetite control hormones before and after the high saturated fat meal challenge at both pre- and post-intervention visits. Appetite control hormones include cholecystokinin (CCK), Peptide YY (PYY), Ghrelin (pg/mL)
Change in fasting and postprandial subjective feelings related to appetite | baseline, 4 weeks
  Visual analog scale ratings of feelings related to appetite before and after the high saturated fat meal challenge, and for the remainder of the day, at both pre- and post- intervention visits. Subjective feelings of hunger, fullness, desire to eat, prospective consumption and a composite appetite score are measured by visual analog scales (mm).
Change in fasting and postprandial plasma Malondialdehyde (MDA) | baseline, 4 weeks
  The concentration of MDA before and after the high saturated fat meal challenge at both pre- and post- intervention visits (nmol/mL).
Change in fasting and postprandial plasma total antioxidant capacity | baseline, 4 weeks
  Total antioxidant capacity before and after the high saturated fat meal challenge at both pre- and post- intervention visits (U/mL).
Change in fasting inflammatory cytokine concentrations | baseline, 4 weeks
  The concentration of interleukin-1 beta, C reactive protein, tumor-necrosis factor-alpha, and interleukin-6 at fasting at both pre-and post-intervention visits (pg/mL).
Change in fasting plasma markers of coagulation potential | baseline, 4 weeks
  The concentration of plasminogen activator inhibitor-1, and tissue factor at fasting for both pre- and post- intervention visits (pg/mL)
Change in fasting and postprandial plasma angiopoietin-like (ANGPTL) proteins | baseline, 4 weeks
  The concentration of ANGPTL 3, ANGPTL 4 and ANGPTL 8 before and after the high saturated fat meal challenge at both pre- and post- intervention visits (ng/mL)
Desaturation index | baseline, 4 weeks
  Measurement of fatty acid concentrations for fasting and post-prandial plasma (ratio of unsaturated to saturated fatty acids)

SECONDARY OUTCOMES:
Change in fasting serum hepatic enzymes | Baseline, 4 weeks
  Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Gamma-Glutamyl Transferase (GGT) (U/L)
Change in fasting serum hepatic proteins | Baseline, 4 weeks
  Total protein and albumin (g/dL)
Change in fasting serum lipoprotein particle numbers | baseline, 4 weeks
  Number of particles of low density lipoproteins (LDL), LDL small, HDL large, LDL medium, lipoprotein (a) (nmol/L)
Change in fasting serum bilirubin | Baseline, 4 weeks
  Total bilirubin, direct bilirubin and indirect bilirubin (mg/dL)
Change in fasting and postprandial plasma insulin concentrations | baseline, 4 weeks
  The concentration of plasma insulin before and after the high saturated fat meal challenge at both pre- and post- intervention visits (uU/mL)
Change in fasting and postprandial plasma glucose concentrations | Baseline, 4 weeks
  The concentration of plasma glucose before and after the high saturated fat meal challenge at both pre- and post- intervention visits (mg/dL)
Change in additional fasting plasma inflammatory cytokine concentrations | baseline, 4 weeks
  The concentration of monocyte chemoattractant protein-1, and interleukin-10, at fasting for both pre- and post-intervention visits (pg/mL)
Change in additional fasting plasma markers of coagulation potential | baseline, 4 weeks
  The concentration of Von Willebrand factor, tissue factor pathway inhibitor, fibrinogen and D-dimer, at fasting for both pre- and post- intervention visits (pg/mL)
Change in acute dietary intake | baseline, 4 weeks
  One-day food logs will be used to record all foods and beverages consumed on testing days
Change in fasting insulin resistance metrics | baseline, 4 weeks
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) and homeostatic model assessment for beta cell function (HOMA-B) will be calculated from fasting insulin and glucose measures before and after the 28-day intervention.

OTHER OUTCOMES:
Change in blood pressure | baseline, 4 weeks
  Systolic and diastolic blood pressure (mmHg)
Change in body weight | baseline, 4 weeks
  body weight (kg)
Change in body composition | baseline, 4 weeks
  DXA will be used to measure body fat percentage (body fat %)
Change in diet composition | baseline, week 2, week 4
  3-day food records will be used to record foods and beverages consumed before and during the 28-day intervention period
Change in fasting tocopherol concentrations | baseline, 4 weeks
  Plasma tocopherol concentrations (ug/mL)
Change in anthropometric circumferences | baseline, 4 weeks
  hip and waist circumferences (cm)
Change in resting metabolic rate | Screening
  Resting metabolic rate (RMR) will be measured for 30 minutes on the TrueOne 2400 (Parvo Medics, Sandy, UT)
Change in Perceived Stress | baseline, 4 weeks
  Perceived Stress Scale will be administered and scored to determine stress levels
Change in anxiety | baseline, 4 weeks
  The State Trait Anxiety Inventory will be administered and scored to determine anxiety levels
Change in self reported physical activity levels | baseline, 2 weeks, 4 weeks
  The International Physical Activity Questionnaire will be used to collect self-reported average physical activity levels (met/min)
Change in Body Mass Index (BMI) | baseline, 4 weeks
  BMI will be calculated based on height and weight measures (kg/m²)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Cooper, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States